CLINICAL TRIAL: NCT01230554
Title: A Study to Assess the Product Performance of a Daily Disposable Contact Lens
Brief Title: Product Performance of a Daily Disposable Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 654
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Myopia
Keywords: contact lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prism I (Experimental): Bausch & Lomb daily disposable cosmetic tint contact lens
  Interventions: Device: Daily disposable cosmetic tint lens

INTERVENTIONS:
Device: Daily disposable cosmetic tint lens — Bausch & Lomb daily disposable cosmetic tint contact lens worn on a daily disposable basis for 1 week.

SUMMARY:
The objective of this one week, single group, bilateral, open-label study is to evaluate the product performance of the Bausch & Lomb daily disposable cosmetic tint contact lens (Test) when worn on a daily disposable basis by adapted current wearers of a marketed opaque tinted soft contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be females of Chinese descent and of legal age and no older than 38. OR subjects that are females of Chinese descent and are at least 15 years of age and less than the legal age must: have a parent/legal guardian provide informed consent.
* Subjects must have clear central corneas and be free of any anterior segment disorders.
* Subjects must be adapted current wearers of marketed opaque tinted soft contact lenses, wear their lenses two days or more per week, and wear a lens in each eye.

Exclusion Criteria:

* Subjects who have worn gas permeable (GP) contact lenses within the last 30 days or have worn polymethylmethacrylate (PMMA) lenses within the last three months.
* Subjects who have any systemic disease affecting ocular health.
* Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Subjects with an active ocular disease or are using any ocular medication.
* Subjects with any scar or neovascularization within the central 4 mm of the cornea.
* Subjects who are aphakic or amblyopic.
* Subjects who have had any corneal surgery (eg, refractive surgery).
* Subjects who currently wear monovision, multifocal, or toric contact lenses.

Ages: 15 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 212 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bausch & Lomb, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prism I
Started | 212
Completed | 209
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Inability to maintain visit schedule | 1

BASELINE CHARACTERISTICS:
Population: Demographics are reported for all eligible, dispensed subjects.
Arm/Group | Prism I
Number analyzed (Participants) | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Market Research Survey
Description: Online subjective assessments that subjects responded to after wearing the study lenses for at least one week. Subjects were asked to rate their overall opinion as: Excellent, Very Good, Good, Fair, or Poor.
Time Frame: 1 week
Population: Subjects who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Prism I
Number analyzed (Participants) | 210
Participants
  Excellent | 10
  Very Good | 91
  Good | 93
  Fair | 16
  Poor | 0

2. Secondary Outcome: Lens Evaluation - Centration
Description: To determine proper lens parameters the lens relationship to the eye was observed using a slit lamp. Lens centration, meaning the lens should provide full corneal coverage, was assessed during the slit lamp evaluation. Findings were reported as: Excellent, Good, Fair, or Poor.
Time Frame: Over all study visits through 1 week
Population: Eligible, dispense eyes with non-missing scores.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Prism I
Number analyzed (Participants) | 212
Number analyzed (eyes) | 424
eyes
  Excellent | 287
  Good | 109
  Fair | 14
  Poor | 14

3. Secondary Outcome: Lens Evaluation - Movement
Description: To determine proper lens parameters the lens relationship to the eye was observed using a slit lamp. Lens movement, meaning the lens should provide discernible movement with:
  * Primary gaze blink
  * Upgaze blink
  * Upgaze lag was assessed during the slit lamp evaluation. Findings were reported as: Adequate, Excessive, Insufficient, Adherence.
Time Frame: Over all study visits through 1 week
Population: Eligible, dispense eyes with non-missing scores.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Prism I
Number analyzed (Participants) | 212
Number analyzed (eyes) | 424
eyes
  Adequate | 246
  Excessive | 0
  Insufficient | 168
  Adherence | 10

4. Secondary Outcome: Visual Acuity - Distance High Contrast logMAR (Logarithm of the Minimum Angle of Resolution) Lens Visual Acuity (VA).
Description: For determination of high contrast VA, the subject was to be seated so that the distance from the subject's eyes to the logMAR chart is 6.5 feet (2.0 meters). The chart should be at eye level for the subject. The logMAR charts have two alternative letter sequences from 28 letters (0.3 logMAR) to 62 letters (-0.3 logMAR). The visual acuity should be measured through the phoropter using the distance refractive correction with the addition of +0.50D to compensate for the reduced test distance of 6.5 feet (2.0 meters).
Time Frame: Over all study visits for 1 week
Population: Eyes with VA results
Measure: Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Prism I
Number analyzed (Participants) | 212
Number analyzed (eyes) | 424
logMAR | 0.012 (0.070)

ADVERSE EVENTS:
Time Frame: Up to 1 week
Description: Adverse events were collected throughout the study.
Arm/Group | Prism I
Serious Adverse Events (participants affected / at risk) | 0/212
Other Adverse Events (participants affected / at risk) | 0/212

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No